CLINICAL TRIAL: NCT01121497
Title: The Effect of Physostigmine on Cognitive Functioning in the Immediate Period After Sedation for Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Prof. Benzion Beilin, Hasharon Hospital, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5759
Record Dates: First submitted 2010-05-09; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-04

CONDITIONS: Cognitive Dysfunction
Keywords: Sedation; Cognitive decline; Physostigmine; Colonoscopy
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Physostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physostigmine (Experimental): Colonoscopy sedation with or without physostigmine
  Interventions: Drug: Physostigmine

INTERVENTIONS:
Drug: Physostigmine — Intravenous bolus of physostigmine 1 mg, 3-5 minutes before completion of the colonoscopy procedure

SUMMARY:
The purpose of this study is to determine whether the administration of physostigmine in combination with sedation for colonoscopy can minimize the cognitive decline at the time of hospital discharge

DETAILED DESCRIPTION:
Physostigmine, a tertiary cholinesterase inhibitor, which prevents the breakdown of ACh by inhibiting the enzyme acetylcholinesterase (AChE), crosses the blood-brain barrier (BBB), and elevates brain ACh levels. Physostigmine has been shown to improve attention, and performance in working memory. It has also been shown to produce analgesia following systemic or central administration.

Patients undergoing colonoscopy under sedation of propofol and fentanyl show cognitive decline in the immediate period following the procedure. In this study, half the patients will receive physostigmine in combination with the sedation, and their cognitive functioning at the time of hospital discharge will be assessed by standard neuropsychological tests, and compared to that of patients without physostigmine.

ELIGIBILITY:
Inclusion Criteria:

* Over18 years old
* ASA I-III
* Fluency in Hebrew, Russian, or Arabic
* Absence of serious hearing or vision impairment

Exclusion Criteria:

* History of head trauma, neurological diseases, alcoholism, drug abuse, consumption of psychotropic drugs or antidepressants
* Heart failure (NYHA > 3)
* Liver failure
* Respiratory problems (asthma, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Cognitive functioning assessed by standard neuropsychological tests | At time of hospital discharge following colonoscopy procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bezion Beilin, MD, Principal Investigator — Hasharon Hospital, Rabin Medical Center
Locations (1):
- Hasharon Hospital, Rabin Medical Center, Petah Tikva, Israel